CLINICAL TRIAL: NCT01250288
Title: Patient Adoption and Use of Health Information Exchange (HIE) Technologies
Brief Title: Usage of Health Information Exchange (HIE) Technologies
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: New York State Department of Health (Other Government); Maimonides Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: C023699-16
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Health Records, Personal
Keywords: Health Information Technology; Health Records, Personal; Hospital Information Systems; Patient Access to Records; Medical Records; Medical Record Systems, Computerized

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Consumers: Consumers (patients or their designated proxies) who have registered to use the personal health management technology platform offered by the Brooklyn Health Information Xchange (BHIX) or Long Island Patient Information Xchange (LIPIX).
  Interventions: Other: Personal Health Management System
- Providers: Providers who are authorized to view the data entered by consumers in either (1) BHIX's personal health management system, along with BHIX health information exchange data; OR LIPIX's secure messaging system (SMS), along with LIPIX health information exchange data.
  Interventions: Other: Personal Health Management System

INTERVENTIONS:
Other: Personal Health Management System — BHIX and LIPIX are offering novel personal health management system to members of its community. These community members, also referred to as consumers, will include patients & their designated proxies. BHIX's system will allow patients to perform various tasks, including, but not limited to, viewing medications, medical allergies and lab results. LIPIX's system is primarily a mechanism forc consumers/patients to communicate directly with their physician through a secure messaging portal. Healthcare providers of these patients, who are affiliated with BHIX, will also be able to view the data entered by consumers in this personal health management system through the RHIO's health information exchange. Thus, the intervention of a personal health management system is being offered to both groups, however in different forms.

SUMMARY:
The purpose of this research study is to describe the usage of consumers and providers when using a novel technology designed to give consumers the ability to manage and access their health information. This is a quantitative descriptive analysis study.

DETAILED DESCRIPTION:
New York State has awarded grants to several regional health information exchange organizations (RHIOs), organizations established to create the technical and policy infrastructure needed to exchange health data between providers, payers, and public health agencies within a particular geographic region, to build an interoperable system for people to manage their own health information. Two of these grant recipients are the Brooklyn Health Information Exchange (BHIX) and Long Island Patient Information Xchange (LIPIX).

Since no off-the shelf technology currently exists to create such a system, BHIX is working with a commercial vendor to develop a unique system that is tailored toward the needs of their consumers and providers, while LIPIX is developing their own unique system in-house. Both BHIX's and LIPIX's interoperable personal health management systems will offer various features to consumers and providers in their community. Consumers may be able to perform tasks such as viewing their lab results, scheduling an appointment, or sending a message directly to their physician through a SMS. Conversely, the PHR can also allow physicians to engage in communications with their patient, release data to their patient(s) (e.g. lab test result); and view patient inputted-data.

The usage patterns of these personal health managements systems is not well understood (Ralson et al., 2009; Kim et al., 2007). Understanding consumers and providers' use of these interoperable systems can help aid in improving current systems and developing future systems.

Specific Aims

The specific aims of this study are to describe the usage of BHIX's and LIPIX's novel interoperable personal health management systems, specifically:

1. To quantify adoption of and frequency of use of novel technological platforms designed to give consumers (patients) access to RHIO-based health information exchange (HIE) data;
2. To quantify usage of HIE-specific data elements within these platforms;
3. To explore associations between usage and user demographics/clinical characteristics;
4. To explore trends in usage over time.

ELIGIBILITY:
Inclusion Criteria:

* Consumers: Consumers (patients or their designated proxies)who are 18 years of age or older and who have registered for either BHIX's personal health record system or LIPIX's secure messaging system.
* Providers: Healthcare Providers who are authorized to view Health Information Exchange data of BHIX or LIPIX.

Exclusion Criteria:

* Anyone that does not fall into the above inclusion category.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consumers (patients and their proxies) and their healthcare providers who are being exposed to a novel interoperable personal health management system in the Brooklyn community.
Sampling Method: Non-Probability Sample
Enrollment: 7800 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Understand Usage Patterns of a Novel Health Information Exchange (HIE) Technology Platform | 1 year
  To describe & quantify the usage of a novel Health Information Exchange (HIE) technology platform in order to understand usage patterns, e.g. frequency of system use; frequency of data element use within theses platforms; associations between usage and user demographics/clinical characteristics. This information can be useful in helping to improve current systems and develop future systems.

SECONDARY OUTCOMES:
Understand Trends in Usage over Time | 1 year
  To describe trends in the usage of a novel HIE technology platform over time. This information can be useful in helping to improve current systems and develop future systems.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica S Ancker, MPH, PhD, Study Chair — Weill Medical College of Cornell University; Rainu Kaushal, MD, MPH, Study Director — Weill Medical College of Cornell University; Melissa C Miller, MPH, Principal Investigator — Weill Medical College of Cornell University; Alison Edwards, MStat, Principal Investigator — Weill Medical College of Cornell University; Yolanda Barron, MS, Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - Brooklyn Health Information Exchange (BHIX), Brooklyn, New York
  - Weill Cornell Medical College, New York, New York
  - Long Island Patient Information Xchange (LIPIX), Rockville Centre, New York